CLINICAL TRIAL: NCT05085028
Title: A Randomised Open-label Phase III Trial of REduced Frequency Pembrolizumab immuNothErapy for First-line Treatment of Patients With Advanced Non-small Cell Lung Cancer (NSCLC) Utilising a Novel Multi-arm Frequency-response Optimisation Design
Brief Title: A Randomised Open-label Phase III Trial of REduced Frequency Pembrolizumab immuNothErapy for First-line Treatment of Patients With Advanced Non-small Cell Lung Cancer (NSCLC)
Acronym: REFINE-Lung
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Medical Research Council (Other Government); University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C/41/2021; 2021-004908-18 (EudraCT Number)
Record Dates: First submitted 2021-10-05; First posted 2021-10-20 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Lung Cancer, Nonsmall Cell
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 6 weekly (Active Comparator): 6 weekly pembrolizumab, 400mg intravenous
  Interventions: Drug: Pembrolizumab 25 MG/ML [Keytruda]
- 9 weekly (Experimental): 9 weekly pembrolizumab, 400mg intravenous
  Interventions: Drug: Pembrolizumab 25 MG/ML [Keytruda]
- 12 weekly (Experimental): 12 weekly pembrolizumab, 400mg intravenous
  Interventions: Drug: Pembrolizumab 25 MG/ML [Keytruda]
- 15 weekly (Experimental): 15 weekly pembrolizumab, 400mg intravenous
  Interventions: Drug: Pembrolizumab 25 MG/ML [Keytruda]
- 18 weekly (Experimental): 18 weekly pembrolizumab, 400mg intravenous
  Interventions: Drug: Pembrolizumab 25 MG/ML [Keytruda]

INTERVENTIONS:
Drug: Pembrolizumab 25 MG/ML [Keytruda] — Pembrolizumab to be given at 400mg intravenous over 5 different frequencies

SUMMARY:
REFINE-lung will test whether reduced pembrolizumab dose frequency after 6 months of standard treatment is safe and effective. Patients treated with 1st line pembrolizumab who are progression free and otherwise planning to continue therapy at 6 months will be initially randomised to control 6 weekly versus interventional 12 weekly therapy. If an interim analysis shows that the 12 weekly treatment is no less effective, subsequent patients will also be randomised to 9, 15 and 18 weekly treatment frequency arms. Patients who progress on a reduced frequency arm will be offered re-escalation to standard 6 weekly therapy.

DETAILED DESCRIPTION:
Immunotherapy with pembrolizumab targeting the T cell inhibitory PD-1 receptor has significantly improved outcomes in advanced non-small cell lung cancer (NSCLC). Approximately 3600 new patients are treated in the 1st line setting per year in England alone and up to 25% remain on 6 weekly pembrolizumab for 2 years. However, pharmacological and clinical trial data suggest current frequent dosing for 2 years result in overtreatment. Indeed, pembrolizumab remains bound to its target receptor for up to 100 days following a single dose and studies in multiple tumour types have found no relationship between dose and patient outcome. Moreover, anti-PD1 treated patients who respond but discontinue therapy either as planned after 2 years, or earlier because of toxicity, can either remain in remission and/or be sensitive to re-challenge with pembrolizumab.

REFINE-lung will test whether reduced pembrolizumab dose frequency (9, 12, 15, 18 weeks) after 6 months of standard treatment is safe and effective.

This UK study represents a unique opportunity to determine whether pembrolizumab dose frequency can be safely reduced in NSCLC, resulting in significant cost benefits to the NHS and globally, in addition to enhanced patient QoL associated with fewer hospital attendances and reduced toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to initiation of any study procedures and willingness and ability to comply with the study schedule
* Any patient ≥18yrs who has received 6 months of pembrolizumab treatment with or without chemotherapy for advanced Non small cell lung cancer who is planned to continue immunotherapy treatment because of continued benefit.

Exclusion Criteria:

* Disease progression or not tolerating treatment at 6 months into therapy
* Clinician does not intend to continue immunotherapy
* Any patient with a synchronous primary cancer. This includes any new cancer diagnoses or relapse of previously treated cancer since starting pembrolizumab treatment.
* Any patient currently receiving an investigational agent and/or using an investigational device or has participated in a study of an investigational agent and/or used an investigational device within 28 days of randomisation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1750 (Estimated)
Dates: Start 2022-06-23 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival at 2 years | 18 months from randomisation
  Survival at 2 years, defined as from commencing pembrolizumab (18 months after randomisation) to death due to any cause or study termination

SECONDARY OUTCOMES:
Overall survival from study entry | 2 years
  Survival, defined as from commencing pembrolizumab (18 months after randomisation) to death due to any cause or study termination
Progression free survival | 2 years
  Progression free survival as assessed by RECIST v1.1, defined as time from study entry to first evidence of disease progression or death due to any cause
Overall response rate | 2 years
  Overall response rate (ORR) as assessed by RECIST v1.1, defined as complete response (CR) or partial response (PR)
Duration of response | 2 years
  Duration of response (DoR) as assessed by RECIST v1.1, defined as time from study entry to change in response from CR or PR to stable disease (SD) or progressive disease (PD)
Incidence of adverse events | 2 years
  Safety and tolerability as assessed by adverse events according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Michael Seckl, Principal Investigator — Imperial College London
Locations (37):
- United Kingdom (37):
  - Royal Bournemouth Hospital, Bournemouth
  - Royal Sussex County Hospital, Brighton
  - Bristol Haematology and Oncology Centre, Bristol
  - Queen's Hospital, Burton-on-Trent
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - East Kent Hospitals University NHS Foundation Trust, Canterbury
  - Velindre Cancer Centre, Cardiff
  - Colchester Hospital, Colchester
  - Royal Derby Hospital, Derby
  - NHS Lothian, Edinburgh
  - Royal Devon and Exeter Hospital, Exeter
  - Beatson West of Scotland Cancer Centre, Glasgow
  - New Victoria Hospital, Glasgow
  - Royal Surrey NHS Foundation Trust, Guildford
  - Calderdale & Huddersfield NHS Foundation Trust, Huddersfield
  - Ipswich Hospital, Ipswich
  - Kettering General Hospital, Kettering
  - NHS Fife, Kirkcaldy
  - Forth Valley Royal Hospital, Larbert
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Leicester Royal Infirmary, Leicester
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Liverpool
  - Guys Hospital, London
  - Imperial College Healthcare NHS Trust, London
  - North Middlesex University Hospital NHS Trust, London
  - St Bartholomew's Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - Northampton General Hospital NHS Trust, Northampton
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Peterborough City Hospital, Peterborough
  - Poole Hospital, Poole
  - Queen's Hospital, Barking Havering and Redbridge University Hospitals NHS Trust, Romford
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - The Royal Marsden NHS Foundation Trust, Sutton
  - Royal Cornwall Hospital, Truro
  - Worthing Hospital, Worthing
  - Yeovil Hospital, Yeovil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ghorani E, Quartagno M, Blackhall F, Gilbert DC, O'Brien M, Ottensmeier C, Pizzo E, Spicer J, Williams A, Badman P, Parmar MKB, Seckl MJ; REFINE-Lung Investigators. REFINE-Lung implements a novel multi-arm randomised trial design to address possible immunotherapy overtreatment. Lancet Oncol. 2023 May;24(5):e219-e227. doi: 10.1016/S1470-2045(23)00095-5. PMID 37142383